CLINICAL TRIAL: NCT05931081
Title: Thermal Imaging in Diagnostics of Chronic Ulcers and in Monitoring Healing of Chronic Ulcers
Acronym: R22108L
Status: Enrolling by invitation | Type: Observational
Sponsor: Tampere University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: R22108L
Record Dates: First submitted 2023-03-23; First posted 2023-07-05 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Chronic Ulcer of Skin

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | US Export: No

INTERVENTIONS:
Device: Thermal imaging in diagnostics of chronic ulcers — atypical: vasculitic or pyoderma gangraenosum ulcers
  Other Names: venous, arterial or mixed ulcers or atypical ulcers

SUMMARY:
Patients with chronic ulcer needing tertiary care referred to the Wound Center of Tampere University Hospital are invited to this study. Patients are treated according to standard treatment practices. The temperature of the lower limbs and ulcer area is measured during visits using the Thermidas Remote thermal imaging system, a CE-marked medical device for measuring and monitoring changes in skin surface temperature non-invasively. The measured temperatures and differences are compared in different ulcer aetiology groups and analyzed whether thermal imaging can be used to distinguish atypical ulcers from vascular ulcers.

Thermal imaging measurements and clinical examinations are repeated to the patients with atypical ulcers during follow-up visits. Monitoring of ulcers will continue until the ulcer has epithelized completely or for up to a year.

DETAILED DESCRIPTION:
4A: Patients with chronic ulcer i.e. venous, arterial or mixed ulcers or atypical (vasculitic or pyoderma gangraenosum) ulcers needing tertiary care referred to the Wound Center of Tampere University Hospital are invited to this study. Aim is to recruit about 20 patients of each group of ulcers. Patients are treated according to standard treatment practices. The temperature of the lower limbs and ulcer area is measured during visits in a standardized measuring environment from both limbs using the Thermidas Remote thermal imaging system (ThRemote 1.3.1, Remote SW with FLIR Inc's series T IR cameras, Thermidas Oy), a CE-marked medical device for measuring and monitoring changes in skin surface temperature non-invasively. The temperature of the ulcer area is compared with the temperature of the corresponding skin area of the other limb and the temperature difference (delta) of the areas is determined. The measured temperatures and differences are compared in different ulcer aetiology groups and analyzed whether thermal imaging can be used to distinguish atypical ulcers from vascular ulcers.

4B: Thermal imaging measurements and clinical examinations are repeated to the patients with atypical ulcers during follow-up visits, and the change in the measurement of temperatures with thermal imaging is compared with the clinician's assessment of the ulcer status (size, ulcer's border activity, necrosis, and pain intensity) and its changes during follow-up visits. Monitoring of ulcers will continue until the ulcer has epithelized completely or for up to a year.

Actual sample size calculations cannot be made, because previous studies on thermal imaging in patients with atypical ulcers have not been published. Based on previous studies, it can be assumed, that statistically significant differences will be obtained between the study groups of approximately 20 subjects. This is a pilot study, and if the study gives promising results, further research will be carried out in the future with more extensive data.

Clinical implication: If thermal imaging is useful in assessing the tendency of ulcer healing, it can be used to optimize the treatment of ulcer patient, such as considering the timing immunosuppressive treatment or skin graft surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic ulcer i.e. venous, arterial or mixed ulcers or atypical (vasculitic or pyoderma gangraenosum) ulcers needing tertiary care referred to the Wound Center of Tampere University Hospital are invited to this study.

Exclusion Criteria:

* Patients with more than one wound etiology in the examined wound (except mixed ulcer) are excluded from the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with chronic ulcer i.e. venous, arterial or mixed ulcers or atypical (vasculitic or pyoderma gangraenosum) ulcers needing tertiary care referred to the Wound Center of Tampere University Hospital are invited to this study.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2025-02-28 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
temperature difference | 1-12 months
  difference of skin temperature between region of an ulcer and healthy skin

SECONDARY OUTCOMES:
healing of an ulcer | 1-12 months
  at least 90% epitelized ulcer

CONTACTS AND LOCATIONS:
Overall Officials: Teija Kimpimäki, Ph.D, Principal Investigator — Tampere University Hospital, University of Tampere
Locations (1):
- Tampere University Hospital, Tampere, Finland

IPD SHARING:
Plan to Share IPD: No